CLINICAL TRIAL: NCT00458887
Title: A Group-Wide, Prospective Study of Ototoxicity Assessment in Children Receiving Cisplatin Chemotherapy
Brief Title: Assessing Ear Damage in Young Cancer Patients Treated With Cisplatin
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACCL05C1; COG-ACCL05C1 (Other: Children's Oncology Group); CDR0000538247 (Other: Clinical Trials.gov)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Ototoxicity; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: ototoxicity; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Ototoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary/Correlative (ototoxicity assessment): Patients undergo hearing tests (conventional, otoscopy, ultrahigh frequency, and otoacoustic emission testing) for management of therapy complications before the first course of planned cisplatin, before each subsequent course of cisplatin, and 4 weeks after the last dose of cisplatin.
  Patients who are scheduled to receive hematopoietic progenitor stem cell transplantation undergo hearing tests for management of therapy complications before the transplantation and 4 weeks after transplantation.
  Interventions: Procedure: management of therapy complications

INTERVENTIONS:
Procedure: management of therapy complications — Undergo hearing tests
  Other Names: complications of therapy, management of

SUMMARY:
RATIONALE: New ways to find out about hearing loss after treatment with chemotherapy may improve the ability to plan cancer treatment and may help patients live more comfortably.

PURPOSE: This clinical trial is assessing ear damage in young cancer patients treated with cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal criteria for determination of ototoxicity in younger cancer patients treated with cisplatin.
* Determine the feasibility of including ultrahigh frequency and evoked otoacoustic emission testing as adjunctive measures of ototoxicity.
* Determine the feasibility and necessity of central review of audiometry data.

OUTLINE: This is a multicenter, prospective, cohort study.

Patients undergo hearing tests (conventional, otoscopy, ultrahigh frequency, and otoacoustic emission testing) before the first course of planned cisplatin, before each subsequent course of cisplatin, and 4 weeks after the last dose of cisplatin.

Patients who are scheduled to receive hematopoietic progenitor stem cell transplantation undergo hearing tests before the transplantation and 4 weeks after transplantation.

PROJECTED ACCRUAL: A total of 282 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planning to undergo treatment with any cisplatin-containing therapeutic regimen for cancer

  * Treatment does not need to be on a COG therapeutic study
* Planning to enroll on clinical trial ACCL0431

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior cisplatin

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients planning to undergo treatment with any cisplatin-containing therapeutic regimen for cancer or planning to enroll on clinical trial ACCL0431
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2007-05; Primary Completion 2015-01 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of patients with ototoxicity according to Common Toxicity Criteria, American-Speech-Language-Hearing Association, and Brock's criteria | Length of study
Proportion of patients who undergo assessments using ultrahigh frequency (UHF) and evoked otoacoustic emission (OAE) testing | Length of study
Proportion of patients with complete standard audiometry data (excluding UHF and OAE evaluations) | Length of Study

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Study Chair — The Hospital for Sick Children
Locations (81):
- United States (73):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - National Naval Medical Center, Bethesda, Maryland
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (7):
  - Children's and Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan